CLINICAL TRIAL: NCT02405338
Title: Dendritic Cell-based Active Immunotherapy of Patients With Acute Myeloid Leukemia Using Autologous Cells Transfected With RNA Encoding Two Different Leukemia-associated Antigens
Brief Title: DC Vaccination for Post-remission Therapy in AML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medigene AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-FDC-001
Record Dates: First submitted 2015-03-24; First posted 2015-04-01 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2019-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WT1/PRAME vaccination (Experimental)
  Interventions: Biological: WT1/PRAME vaccination

INTERVENTIONS:
Biological: WT1/PRAME vaccination

SUMMARY:
This is a multi-centre, open label, prospective, non-randomized phase I/II trial in 20 patients including a safety-run in phase I part comprising 6 patients.

Trial subjects will receive repeated immunotherapies with autologous Dendritic Cells (DCs), presenting two leukemia-associated antigens.

DETAILED DESCRIPTION:
20 patients with AML who are in remission (ELN criteria by Döhner et al 2017) receive WT1/PRAME autologous DC vaccine by intradermal injection once per week during the first 4 weeks and 1 per month thereafter for 23 consecutive months.

Primary objective is to assess the safety and tolerability of the DC vaccine in the aforementioned population and the feasibility.

Secondary objectives include evaluation of clinical response and exploratory immune monitoring assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Myeloid Leukemia (AML)
* Age 18 - 75 years
* Morphologic remission (CR) with or without hematological recovery (CRi) following induction chemotherapy
* WT1 with or without PRAME positivity by qPCR
* Negative pregnancy test in women of childbearing potential (within 7 days before the first vaccination). Women of childbearing potential and sexually active male participants must use reliable methods of contraception during the whole treatment period and 3 months after the last trial drug dose
* Negative HIV 1 and 2 test, Hepatitis B and C test and negative Syphilis test at screening
* Informed consent signed prior to any trial related activities

Exclusion Criteria:

* Patients suitable for allogeneic stem cell transplantation
* AML M3 (acute promyelocytic leukemia)
* Patients not in complete remission (CR or CRi), bone marrow blast count ≥ 5 %
* Active immunodeficiency syndromes
* Concurrent active second malignancy other than non-melanoma skin cancers
* Clinically relevant autoimmune disease
* Prior immunotherapy
* Severe organ dysfunction precluding the apheresis procedure:
* Creatinine > 200 mmol/l
* Bilirubin, ALAT and ASAT > 3 x upper normal limit
* Respiratory insufficiency with pO2 < 60 mmHg
* Clinically relevant coronary heart disease of ventricular arrhythmia, congestive heart failure > grade II NYHA
* Recent cerebral hemorrhage
* Known allergies to substances used in the generation of DCs
* Other severe acute or chronic medical psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or the administration of the investigational product
* Use of corticosteroids
* Active CMV infection (Antibody-positivity due to previous, now inactive infection is accepted)
* Inability to comply with the trial protocol
* Participation in other clinical trials that, according to the investigator's discretion, may interfere with this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in whom treatment with the scheduled number of immunotherapies is feasible | 2 years
Percentage of grade I/II, grade III/IV and grade ≥III toxicities in patients having received at least 1 immunotherapy | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Relapse/Progression free survival | 2 years
Time to progression (TTP). | 2 years
Control of minimal residual disease (MRD) | 2 years
ECOG performance status | 2 years
Cellular immune responses to applied antigens | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yngvar Fløisand, Principal Investigator — Oslo University Hospital, Rikshospitalet Department of Hematology
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway